CLINICAL TRIAL: NCT01822652
Title: Autologous Activated T-Cells Transduced with a 3rd Generation GD-2 Chimeric Antigen Receptor and ICaspase9 Safety Switch Administered to Patients with Relapsed or Refractory Neuroblastoma (GRAIN)
Brief Title: 3rd Generation GD-2 Chimeric Antigen Receptor and ICaspase Suicide Safety Switch, Neuroblastoma, GRAIN
Acronym: GRAIN
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); Solving Kids' Cancer (Other); The Evan Foundation (Other); National Cancer Institute (NCI) (NIH); Kids Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Andras Heczey, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-31493 GRAIN; P01CA094237 (NIH)
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Solid tumor; Neuroblastoma-specific immunotherapy targeting GD2; CAR T cells; Gene Therapy; Relapsed; Refractory
MeSH Terms: conditions — Neuroblastoma; Recurrence | interventions — Cyclophosphamide; fludarabine phosphate; fludarabine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- iC9-GD2 T Cells - fresh - CLOSED (Experimental): The cells will be given IV over 5-10 minutes. There is a possibility for additional doses of iC9-GD2 T cells.
  Interventions: Genetic: iC9-GD2 T Cells - fresh
- iC9-GD2 T Cells - frozen - CLOSED (Experimental): The cells will be given IV over 5-10 minutes. There is a possibility for additional doses of iC9-GD2 T cells.
  Interventions: Genetic: iC9-GD2 T Cells - frozen
- iC9-GD2 T cells,Cytoxan,Fludara,Keytruda (Experimental): Fresh T cells will be given IV over 5-10 mins. There is a possibility for additional doses of iC9-GD2 T cells.
  Interventions: Drug: Cytoxan; Drug: Fludara; Drug: Keytruda; Genetic: iC9-GD2 T cells

INTERVENTIONS:
Genetic: iC9-GD2 T Cells - frozen — Subjects will receive the iC9-GD2 T cells through an IV over 5 to 10 minutes.
  Subjects will receive one of the following dose levels (cells/m2):
  * Dose Level 1 = 1 x 10^7
  * Dose Level 2 = 1 x 10^8
  * Dose Level 3 = 2 x 10^8
  Six weeks after the infusion, patients will have a disease re-evaluation. If the disease has not gotten worse AND they have not had a severe side effect caused by the infusion of the iC9-GD2 T cells, the subject may be eligible to receive up to 2 additional doses of T cells. Each dose will be at the same dose level as the first infusion, if available, and separated by at least 6 weeks.
  Arms: iC9-GD2 T Cells - frozen - CLOSED
Genetic: iC9-GD2 T Cells - fresh — For subjects who will receive a fresh T cell product:
  * Dose Level 1 = 1 x 10^8
  * Dose Level 2 = 1.5 x 10^8
  * Dose Level 3 = 2 x 10^8
  Six weeks after the infusion, patients will have a disease re-evaluation. If the disease has not gotten worse AND they have not had a severe side effect caused by the infusion of the iC9-GD2 T cells, the subject may be eligible to receive up to 2 additional doses of T cells. Each dose will be at the same dose level as the first infusion, if available, and separated by at least 6 weeks.
  Arms: iC9-GD2 T Cells - fresh - CLOSED
Drug: Cytoxan — Cyclophosphamide (500 mg/m2/day x 2 days, for patients <12 kg = 16.7 mg/kg/day x 2 days)
  Other Names: Cyclophosphamide
  Arms: iC9-GD2 T cells,Cytoxan,Fludara,Keytruda
Drug: Fludara — Fludarabine (30 mg/m2/day x 3 days, for patients <12 kg = 1 mg/kg/day x 3 days)
  Other Names: Fludarabine
  Arms: iC9-GD2 T cells,Cytoxan,Fludara,Keytruda
Drug: Keytruda — Pembrolizumab (2 mg/kg on Day -1 and on Day 21).
  Other Names: Pembrolizumab
  Arms: iC9-GD2 T cells,Cytoxan,Fludara,Keytruda
Genetic: iC9-GD2 T cells — For subjects who will receive a fresh T cell product:
  * Dose Level 1 = 1.5 x 10^8
  * Dose Level 2 = 2 x 10^8
  Six weeks after the infusion, patients will have a disease re-evaluation. If the disease has not gotten worse AND they have not had a severe side effect caused by the infusion of the iC9-GD2 T cells, the subject may be eligible to receive up to 2 additional doses of T cells. Each dose will be at the same dose level as the first infusion, if available, and separated by at least 6 weeks.
  Arms: iC9-GD2 T cells,Cytoxan,Fludara,Keytruda

SUMMARY:
Subjects that have relapsed or refractory neuroblastoma are invited to take part in this gene transfer research study.

We have found from previous research that we can put a new gene called a chimeric antigen receptor (CAR) into T cells that will make them recognize neuroblastoma cells and kill them. In a previous clinical trial, we used a CAR that recognizes GD2, a protein found on almost all neuroblastoma cells (GD2-CAR). We put this gene into T cells and gave them back to patients that had neuroblastoma. The infusions were safe and in patients with disease at the time of their infusion, the time to progression was longer if we could find GD2 T cells in their blood for more than 6 weeks. Because of this, we think that if T cells are able to last longer, they may have a better chance of killing neuroblastoma tumor cells.

Therefore, in this study we will add new genes to the GD2 T cells that can cause the cells to live longer. These new genes are called CD28 and OX40. The purpose of this study will be to determine the highest dose of iC9-GD2-CD28-OX40 (iC9-GD2) T cells that can safely be given to patients with relapsed/refractory neuroblastoma.

In other clinical studies using T cells, some investigators found that giving chemotherapy before the T cell infusion can improve the amount of time the T cells stay in the body and therefore the effect the T cells can have. This is called lymphodepletion and we think that it will allow the T cells we infuse to expand and stay longer in the body, and potentially kill cancer cells more effectively.

The chemotherapy we will use for lymphodepletion is a combination of cyclophosphamide and fludarabine.

Additionally, to effectively kill the tumor cells, it is important that the T cells are able to survive and expand in the tumor. Recent studies have shown that solid tumors release a substance (PD1) that can inhibit T cells after they arrive into the tumor tissue. In an attempt to overcome the effect of PD1 in neuroblastoma we will also give a medication called pembrolizumab.

DETAILED DESCRIPTION:
We will make iC9-GD2 T cells by infecting normal T cells with a retroviral vector containing the iC9-GD2 gene. After the new gene has been put into the T cells, the cells will be tested to make sure that they kill GD2-positive neuroblastoma cells and then will be either given fresh or frozen until the patient is ready for their infusion.

First, patients will receive cyclophosphamide and fludarabine intravenously (through a needle inserted into a vein or your port-a-cath) for 2 days and then fludarabine alone for one day (Day -4, -3,-2). On the next day (Day -1) patients will receive the drug called pembrolizumab intravenously. Finally on Day 0 patients will be given an infusion of iC9 GD2 T cells into the vein through an IV line at the assigned dose.

The iC9-GD2 T cell infusion will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital. The infusion will take between 5 and 10 minutes. Patients may need to stay in Houston for up to 4 weeks after the infusion so we can monitor them for side effects.

On Day 21 (at the time of the week 3 visit), if the treatment was well tolerated, patients will receive another dose of pembrolizumab intravenously.

There will be follow-up visits every 1-2 weeks during the first 2 months and then they will be spaced out over a total of 15 years. Because the cells are modified with a new gene we must follow patients for at least 15 years to see if there are any long term side effects of gene transfer. During the visits, we will see how the patients are doing and during certain time points we will obtain extra blood samples to learn more about the way the iC9-GD2 T cells are working and how long they last in the body.

After disease re-evaluation, if disease has not gotten worse, or if in the future it seems that patient might benefit and they have not had a severe side effect caused by the infusion of their iC9-GD2 T cells, patients may be eligible to receive up to 2 additional doses of their T cells. Each dose will be at the same dose level as their first infusion and separated by at least 6 weeks such that we can make sure patients have no severe side effects between infusions. If patients receive additional doses of iC9-GD2 T-cells, they may need to stay in Houston for up to 4 weeks after the infusion as well so we can monitor them for side effects. If there were no severe side effects from pembrolizumab, patients will receive pembrolizumab again with the iC9 GD2 T cells on the day before the T cell injection and 21 days after the T cells.

ELIGIBILITY:
Inclusion Criteria:

PROCUREMENT

* High risk neuroblastoma with persistent or relapsed disease
* Life expectancy of at least 12 weeks
* Karnofsky/Lansky score of 60% or greater
* Absence of HAMA prior to enrollment (only in patients that have been previously treated with murine antibodies)
* Informed consent and assent (as applicable) obtained from parent/guardian and child

TREATMENT:

* High risk neuroblastoma with persistent or relapsed disease
* Life expectancy of at least 12 weeks
* Karnofsky/Lansky score of 60% or greater
* Patients must have an ANC greater than or equal to 500, platelet count greater than or equal to 20,000
* Pulse Ox greater than or equal to 90% on room air
* AST and ALT less than 5 times the upper limit of normal
* Total bilirubin less than 3 times the upper limit of normal
* Serum creatinine less than 3 times upper limit of normal. Creatinine clearance is needed for patients with creatinine greater than 1.5 times upper limit of normal
* TSH normal for age. Patients using thyroid medication to facilitate a euthyroid state must be on a stable dose for at least 1 month prior to planned infusion
* Recovered from acute effects of all prior chemotherapy. If some effects of therapy have become chronic (i.e., treatment associated thrombocytopenia), the patient must be clinically stable and meet all other eligibility criteria
* Absence of human anti-mouse antibodies (HAMA) prior to enrollment for patients who have received prior therapy with murine antibodies
* Patients must have autologous transduced activated T-cells with greater than or equal to 20% expression of GD2
* Pembrolizumab available for infusion
* Informed consent and assent (as applicable) obtained from parent/guardian and child

Exclusion Criteria:

PROCUREMENT:

* Rapidly progressive disease
* History of hypersensitivity to murine protein containing products

TREATMENT:

* Rapidly progressive disease
* Currently receiving other investigational drugs
* History of hypersensitivity to murine protein containing products
* History of cardiomegaly or bilateral pulmonary infiltrates on chest radiograph or CT. However, patients with cardiomegaly on imaging may be enrolled if they have an assessment of cardiac function (i.e., ECHO or MUGA) within 3 weeks of starting protocol therapy that is within normal limits. Additionally, patients with bilateral pulmonary infiltrates on imaging may be enrolled if the lesions are not consistent with active neuroblastoma (i.e., negative on functional imaging with PET or MIBG, or by pathologic assessment).
* Evidence of tumor potentially causing airway obstruction
* Patients who are pregnant, lactating, or unwilling to use birth control
* Patients currently receiving immunosuppressive drugs such as corticosteroids, tacrolimus or cyclosporine
* Patients previously experienced severe toxicity from cyclophosphamide or fludarabine
* Severe previous toxicity from pembrolizumab or other PD-1 targeted antibody

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities at 6 weeks post T cell infusion | 6 weeks after infusion of the last dose of iC9-GD2 T cells to all patients on the study
  We will measure and assess the adverse events to find the maximum tolerated dose of iC9-GD2 T cells and the safety profile of iC9-GD2 T cells.

SECONDARY OUTCOMES:
To evaluate the expansion and persistence of 3rd generation iC9-GD2 T cells | 15 years
  We will determine the expansion and functional persistence of iC9-GD2 T cells in the peripheral blood of patients using transgene detection by quantitative real-time PCR and response of transgenic cells to tumor antigen and to dimerizing drug in vitro.
Time to progression of disease | 15 years
  To describe the overall response rate and disease-free survival.
Change in serum cytokine and chemokine levels | 15 years
  The changes in patients' serum cytokine and chemokine levels after iC9-GD2 T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Andras A. Heczey, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas